CLINICAL TRIAL: NCT01996969
Title: Identification of Predictive Biomarker of Regorafenib in Refractory Colorectal Cancer: A Prospective Explorative Study
Brief Title: Identification of Predictive Biomarker of Regorafenib in Refractory Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Tae-You Kim, M.D., Ph.D, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Regorafenib biomarker
Record Dates: First submitted 2013-10-24; First posted 2013-11-27 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; refractory; regorafenib; biomarker; gene sequencing
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Other): This study is a single arm study with biomarker analysis
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib will be given 160mg once daily for 3 weeks, followed by a 1 week rest. Treatment will be continued until disease progression or unacceptable toxicity occurs. Response evaluation (CT scans) will be performed every 2 cycles.

SUMMARY:
Regorafenib is a valuable treatment option for metastatic colorectal cancer patients who have progressed after prior standard treatments. Prior progression-free survival data suggest that there could be a distinct subgroup of patients that may benefit from regorafenib. The aim of this study is to identify predictive biomarker of regorafenib in terms of its efficacy.

DETAILED DESCRIPTION:
Regorafenib is a multi-tyrosine kinase inhibitor which has been shown to increase survival in metastatic colorectal cancer patients who have progressed after prior standard treatments. Progression-free survival data suggest that there could be a distinct subgroup of patients that may benefit from regorafenib. Therefore, it would be important to identify predictive biomarker of efficacy of regorafenib. Considering that regorafenib is a multi-tyrosine kinase inhibitor, comprehensive approach is required to discover predictive biomarker.

NGS-based sequencing allows generating large amount of data regarding multiple genes and multiple genetic alterations within a single experiment. Also, it requires less amount of DNA or tissue and cost compared to currently used individual gene testing techniques such as direct sequencing or FISH. Moreover, superior sensitivity over Sanger sequencing can be obtained by increasing coverage depth, especially in cases with low tumor purity. Wide range of genes targeted by regorafenib and genes in the major oncogenic pathway of colorectal cancer influenced by regorafenib can be efficiently assessed using NGS-based sequencing.

The aim of this study is to identify predictive biomarker of efficacy of regorafeinib in metastatic, refractory colorectal cancer patients using NGS technology.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any study-specific procedures.
2. Age ≥ 20
3. Pathologically confirmed metastatic adenocarcinoma of colon or rectum
4. Failure of standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan. Failure is defined as progression during or within 3 months following the last administration of therapy. Patients who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent before progression of disease will also be allowed into the study. Patients treated with oxaliplatin in an adjuvant setting who have progressed during or within 6 months of completion of adjuvant therapy are regarded as failure of oxaliplatin. Patients may or may not have received bevacizumab or cetuximab.
5. Measurable or nonmeasurable disease according to RECIST criteria, version 1.1.
6. Adequate tissue for gene sequencing (surgical FFPE specimen or fresh-frozen biopsy specimen)
7. ECOG PS 0 or 1
8. Life expectancy of at least 3 months
9. Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 14 days of starting to study treatment

   * Total bilirubin ≤1.5 × ULN
   * Alanine aminotransferase and aspartate aminotransferase ≤2 × ULN (≤5 × ULN for patients with liver involvement of cancer)
   * Amylase and lipase ≤1.5 × ULN
   * Serum creatinine ≤1.5 × ULN
   * Glomerular filtration rate ≥30 ml/min/1.73 m2 according to the Modified Diet in Renal Disease abbreviated formula
   * International normalised ratio (INR) and partial thromboplastin time (PTT) ≤1.5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of an underlying abnormality in coagulation parameters exists.
   * Platelet count ≥100,000/mm3, haemoglobin >9 g/dl, absolute neutrophil count >1,500/mm3
   * Alkaline phosphatase limit ≤2.5 × ULN (≤5 × ULN for patients with liver involvement of their cancer)

Exclusion Criteria:

1. Prior treatment with regorafenib
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
3. Pregnancy or breast-feeding. Women of childbearing potential must have a negative pregnancy test performed a maximum of 7 days before start of treatment
4. Congestive heart failure of NYHA class 2 or worse
5. Unstable angina, new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study drug
6. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
7. Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic >90 mmHg despite optimal medical management)
8. Arterial or venous thrombotic or embolic events within the 6 months before start of study medication
9. Ongoing infection higher than NCI-CTCAE v4.0 grade 2
10. Known history of HIV infection
11. Active hepatitis B or C virus infection
12. Seizure disorder requiring medication
13. Symptomatic metastatic brain or meningeal tumors
14. History of organ allograft
15. Non-healing wound, ulcer, or bone fracture
16. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
17. Persistent proteinuria of NCI-CTCAE v4.0 grade 3 or higher
18. Inability to swallow oral medications
19. Any malabsorption condition
20. Unresolved toxicity higher than NCI-CTCAE v4.0 grade 1 attributed to any prior therapy/procedure, excluding alopecia and oxaliplatin-induced neurotoxicity of grade 2 or less

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Predictive biomarker in terms of disease control rate | 1 year
  This study aims at identifying potential molecular subgroup of colorectal cancer that may benefit from regorafenib treatment in terms of disease control rate.

SECONDARY OUTCOMES:
Disease control rate | 1 year
  Disease control rate in all treated population
Progression-free survival | 1 year
  Progression-free survival in all treated population
Overall survival | 1 year
  Overall survival in all treated population
number of participants with adverse events | 1 year
  adverse events according to NCI-CTCAE v.4.0
Progression-free survival according to biomarker status | 1 year
  Progression-free survivals will be compared according to biomarker status
Overall survival according to biomarker status | 1 year
  Overall survivals will be compared according to biomarker status
Assessment of adequate response evaluation modality after regorafenib treatment | 1 year
  Changes in size, CT attenuation (HFU) and PET metabolism (SUV) will be evaluated and assessed in relation to survival outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Tae-You Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital; Sae-Won Han, M.D.,Ph.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea